CLINICAL TRIAL: NCT04847804
Title: Large-scale Population Screening of Pooled Viral Nucleic Acid Samples Using Concurrent Isothermal Amplification and Electrochemical Detection for Novel Infectious Diseases on a Disposable Chip
Brief Title: Large-scale COVID-19 Population Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Kong University of Science and Technology (Other)
Collaborators: Chinese University of Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, I-Ming Hsing, Professor, Department of Chemical and Biological Engineering, Hong Kong University of Science and Technology
Other Study IDs: CRE2021.188
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: COVID-19; Population screening
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — nasopharyngeal swab, deep throat saliva, and/or mouth gargle sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive case: The sample will be tested by microfluidic device and shows positive
- Negative control: The sample will be tested by microfluidic device and shows negative

SUMMARY:
Infectious diseases pose a threat to the life of individuals worldwide. The pandemic has highlighted the need to develop an innovative and cost- effective large population-based screening methodology. The investigators propose a two-fold improvement barcode-labeled testing strategy specifically for pooled samples. This platform combines isothermal amplification and real-time electrochemical detection; electroactive modified loop probes will be used in the amplification step for barcode readout. This method enables four samples pooled detection at the same time. This platform will be integrated into a disposable microfluidic chip that allows minimal human intervention during the process to realize a massively parallel screening platform for infectious disease pathogens.

Objectives

1. To develop a sensing method for concurrent electrochemical-tag coded isothermal amplification and real-time electrochemical detection;
2. To design a molecular strategy to barcode four individual samples so that they can be pooled together and to simultaneously amplify and identify a positive individual, if any, from the pooled sample.
3. To fabricate a microfluidic device integrating the sample processor and barcoding module with the nucleic acid amplification and detection step for large-scale population screening of up to 100 individuals.
4. To validate the performance of the prototype using clinical specimens and benchmark it against the detection data from commercially available testing equipment.

DETAILED DESCRIPTION:
Rapid host-to-host transmissions coupled with the ease of international travel has led to epidemics such as H5N1, H5N5, SARS, and, most recently, the COVID-19 pandemic. Traditional epidemic control measures, such as contact tracing and physical isolation, are paramount to mitigate the extent of disease spread at the early stage of the pandemic and these strategies depend on the accuracy and speed of diagnosing suspected patients.

Now the gold standard for pathogen detection is nucleic acid detection via polymerase chain reaction (PCR). However, this strategy is limited by the turnaround time, expensive PCR machine, and potential number of infections. Thus, other isothermal amplification methods are often used to circumvent the need for extra instrumentation and speed up the whole detection procedure.

One approach to improve infectious disease screening efficiency is the popular Dorfman testing, where samples are pooled together and tested at the same time to reduce the total number of tests performed. However, the Dorfman testing is limited to low prevalence population and has reduced sensitivity; Barcoding strategy has also been introduced to solve pooling sample test. In 2020, Schmid-Burk and his colleagues combined LAMP and barcoding which successfully developed COVID-19 from 100,000 pooled samples. However, the need of a expensive next-generation sequencer limits its widespread use.

Methods

The proposed platform aims at development of a multistep process in one device, and the capability of identifying the source of positive signals from pooled samples. The proposed design will take advantage of a barcoding strategy to tag multiple sources of analytes prior to pooling, a combination of isothermal amplification and sequence-specific electrochemical detection, and the integration of several steps in one simple device. The research project methodology will be divided into three parts.

(i) To develop an isothermal amplification method and real-time detection using electroactive-labelled loop oligonucleotide probes

The investigators have recently conceptualized a method, for which the investigators have filed a US provisional patent protection. This new technique performs the isothermal amplification and electrochemical detection of amplicons simultaneously based on Loop-mediated isothermal amplification (LAMP). The proposed scheme involves a one-pot amplification and detection system in which an electrochemical reporter is attached to one of the primers and a nicking enzyme is added to cleave the reporter only when amplification occurs. In one reaction, a template DNA is designed to have two pairs of primer binding sites: an outer pair of forward and backward primers (FP and BP) and an inner pair of primers, namely, an electrochemically labeled loop probe (LP) and an assistant probe (AP). The FP and LP bind to the same strand of the double-stranded DNA (dsDNA) template while the BP and AP bind to the opposite strand. The LP contains an electroactive label at the 5' end and a 3' overhanging segment complementary to the target DNA sequence. The stem region contains the recognition sequence of a nicking enzyme, but a mismatch is introduced to the last nucleotide so that it will not be cleaved without the presence of the target DNA. The start of the reaction is similar to ordinary LAMP, a double-loop amplicon can be produced, and the reaction can come into the double loop amplification stage. Each of the double-loop amplicons can be regarded as a signal amplification unit. Once the labeled LP is combined with the amplicon and form a cleavage site that can be recognized by the nick enzyme, an electroactive label can be released, and an electrochemical signal will be generated. The preliminary results indicate that the strategy is able to detect up to 0.1 fg/μL, corresponding to around 10 copies/μL of the input DNA, by using a methylene blue electroactive reporter on four-array screen-printed carbon electrodes (SPCEs) within 30 min. The succeeding steps include incorporating a reverse transcription step for the detection of RNA samples and testing the system in complex matrices to mimic actual biological fluids.

(ii) To design a molecular strategy to barcode four individual samples so that they can be pooled together and to simultaneously amplify and identify the positive individual, if any, from the pooled sample.

By designing four barcode sequences, the investigators are able to construct tagged cDNA products through reverse transcription by BST enzyme. Thermolabile exonuclease I is added to digest unreacted single strand barcode primers. In addition, the cDNA-RNA duplex product is digested by RNase H to yield a single-stranded cDNA (ID-template).The pooled mixture of ID-templates is amplified through the same process described in the previous section. Only those samples with the RNA virus will generate positive electrochemical signals.

In this part, the investigators will use synthesis virus RNA or commercial extracted virus total RNA as a detection template. The spiked samples can be mocked by mixing with human deep throat saliva or nasopharyngeal swabs from healthy volunteers.

(iii) To fabricate a microfluidic device to integrate the sample processor and barcoding module with the nucleic acid amplification and detection step for large-scale population screening

In this project, the investigators design a simple and easy-to-use microfluidic pen-like device that integrates the steps of sample preparation, barcoding, and amplification and detection. It uses piston propulsion to provide power to push the sample into different chambers. First, the mock samples are added into a sample loading chamber where the lysis buffer is stored. A mixture of surfactin, SDS, and ethanol allows the rapid extraction of viral nucleic acid, which is then injected down to the identification chamber containing the freeze-dried BST polymerase and ID-tag primer mixture. The temperature will remain at 37 °C-50°C for reverse transcription. Then, the sample is injected to the chamber containing thermolabile exonuclease I. The heating block is then set to 65 °C for 5 min to deactivate the enzyme. Thereafter, the four samples are pooled together and injected into an electrochemical detection chip below the microfluidic pen. Each chip contains four sets of primers and LPs with different electroactive reporters with non-overlapping redox potentials to trigger the amplification reaction in the presence of respective participant's ID sequences.

The detection chamber sits atop a multichannel electrochemical workstation, which consists of a connection port between the electrochemical sensor and detector, a circuit board, and a power line for external display. The circuit board is mainly composed of a microcontroller unit, a digital-to-analog converter, and a potentiostat module to allow for differential pulse voltammetry analysis and simultaneously obtain the signals from an array of electrodes and thereby detect a total of 100 samples.

(iv) To validate the performance of the prototype using a clinical specimen and benchmark it against the detection data from commercially available testing equipment.

The proposed method of pooled sample testing will be compared with the gold standard RT-PCR test in terms of sensitivity, specificity, positive predictive value, negative predictive value, and accuracy. After demonstrating the validity of the results obtained from the proposed pooling strategy, the investigators will then explore the possibility of using saliva and mouth gargle samples in lieu of the nasopharyngeal swabs. Patients will be recruited from the Prince of Wales Hospital for collection of respiratory samples to determine the accuracy of this device.

A. Study procedures

1. Participants' medical records to collect clinical data, including age, sex, number of days after the onset of symptoms, epidemiological exposure to people with confirmed COVID-19 disease, severity (mild, moderate, severe, or critical), and the presence of comorbidities will be reviewed.
2. SARS-CoV-2 PCR results of the participants from hospital electronic record will be retrieved.
3. Nasopharyngeal swab, deep throat saliva, and/or mouth gargle sample from each recruited patient will be collected.

B. Laboratory procedures and data analyses

1. Sample preparation The samples collected from the 200 patients will firstly be divided for two sets with similar prevalence, and each sample size is 100. The first set 100 samples will be extracted by using commercial viral RNA extraction kits provided by HKUST, and then be stored for further RT-qPCR analysis and the LAMP-based method verification.
2. RT-qPCR assay To prepare RT-qPCR result as the reference, the extracted samples from mentioned above will be analyzed using RT-qPCR for the qualitative and quantitative detection of nucleic acid from the SARS-CoV-2, and a negative, a positive and a blank control experiment should be included. The cycle thresholds (Ct) values, qualitative and quantitative results of each sample will be recorded. The RT-qPCR procedures will be followed by existing CDC-recommended guidelines. The qPCR primer and Taqman probe sets, and SARS-CoV-2 RNA standard reference will be provided by HKUST.
3. Pooled sample experiments The second set 100 inactivated samples will be divided into 25 groups randomly (each for 4 samples), and the investigators will perform SARS-CoV-2 group testing for the 25 pools using the microfluidic device developed above with HKUST researchers. Based on the RT-qPCR results, the sensitivity, specificity, and positive and negative predictive values will be calculated for further data analysis by HKUST.

Study conduct

This study will be conducted in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at the Prince of Wales Hospital who have received testing for SARS-CoV-2 PCR
* Age 18 years or above

Exclusion Criteria:

* Mentally incompetent to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized at the Prince of Wales Hospital who have received testing for SARS-CoV-2 PCR
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic test | through study completion, an average of 3 years
  The sensitivity, specificity, and positive and negative predictive values will be calculated for futher data analysis

CONTACTS AND LOCATIONS:
Overall Officials: I-Ming HSING, Principal Investigator — Hong Kong University of Sciences and Technology
Locations (3):
- Hong Kong (3):
  - The Hong Kong University of Sciences and Technology, Sai Kung
  - Chinese University of Hong Kong, Shatin
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollingsworth TD, Ferguson NM, Anderson RM. Frequent travelers and rate of spread of epidemics. Emerg Infect Dis. 2007 Sep;13(9):1288-94. doi: 10.3201/eid1309.070081. PMID 18252097
- [Background] Hufnagel L, Brockmann D, Geisel T. Forecast and control of epidemics in a globalized world. Proc Natl Acad Sci U S A. 2004 Oct 19;101(42):15124-9. doi: 10.1073/pnas.0308344101. Epub 2004 Oct 11. PMID 15477600
- [Background] Ferretti L, Wymant C, Kendall M, Zhao L, Nurtay A, Abeler-Dorner L, Parker M, Bonsall D, Fraser C. Quantifying SARS-CoV-2 transmission suggests epidemic control with digital contact tracing. Science. 2020 May 8;368(6491):eabb6936. doi: 10.1126/science.abb6936. Epub 2020 Mar 31. PMID 32234805
- [Background] Shears P. Emerging and reemerging infections in africa: the need for improved laboratory services and disease surveillance. Microbes Infect. 2000 Apr;2(5):489-95. doi: 10.1016/s1286-4579(00)00309-9. PMID 10865194
- [Background] Lazcka O, Del Campo FJ, Munoz FX. Pathogen detection: a perspective of traditional methods and biosensors. Biosens Bioelectron. 2007 Feb 15;22(7):1205-17. doi: 10.1016/j.bios.2006.06.036. Epub 2006 Aug 28. PMID 16934970
- [Background] Jani IV, Janossy G, Brown DW, Mandy F. Multiplexed immunoassays by flow cytometry for diagnosis and surveillance of infectious diseases in resource-poor settings. Lancet Infect Dis. 2002 Apr;2(4):243-50. doi: 10.1016/s1473-3099(02)00242-6. PMID 11937424
- [Background] R. Dorfman, The Detection of Defective Members of Large Populations, Ann. Math. Stat. 14 (1943) 436-440.
- [Background] J.L. Schmid-burgk, D. Li, D. Feldman, J. Strecker, B. Cleary, A. Regev, LAMP-Seq : Population-Scale COVID-19 Diagnostics Using a Compressed Barcode Space, BioRxiv. (2020).